CLINICAL TRIAL: NCT02869152
Title: Novel Sentinel Lymph Node Mapping Technique in Early Stage Rectal Cancer
Brief Title: Sentinel Lymph Node Mapping in Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Traci Hedrick, MD, Assistant Professor of Surgery, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19120
Record Dates: First submitted 2016-07-14; First posted 2016-08-16 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Rectal Neoplasms
Keywords: sentinel lymph node; lymphatic mapping; rectal tumor; rectal cancer; early stage
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraoperative sentinel lymph node mapping (Experimental): Subjects will come to the OR and undergo a flexible sigmoidoscopy after induction of anesthesia and receive separate endoscopic injections of Spot (up to 5 cc), 99mTc-sulfur colloid (up to 0.5 mCi), and Indocyanine green (ICG) (1 ml). Patient will undergo the standard transanal endoscopic surgery (TES) to remove the rectal neoplasm, exposing the lymph node basin. The sentinel node(s) will be identified using a combination of the gamma probe and fluorescence imaging endoscopically, dissected out, and removed through a transanal approach.
  Interventions: Other: Endoscopic injection of 99mTc-sulfur colloid; Other: Endoscopic injection of ICG; Other: Endoscopic injection of Spot; Procedure: Flexible sigmoidoscopy; Procedure: Endoscopic NIR imaging and gamma probe; Procedure: Dissection of sentinel lymph node(s)

INTERVENTIONS:
Other: Endoscopic injection of 99mTc-sulfur colloid — Radiotracer injection around the rectal tumor for SLN mapping with gamma probe
Other: Endoscopic injection of ICG — Dye injection around the rectal tumor for SLN mapping with NIR imaging.
Other: Endoscopic injection of Spot — Dye injection for tattooing rectal tumor prior to surgical resection.
Procedure: Flexible sigmoidoscopy — Flexible sigmoidoscopy prior to surgery to facilitate endoscopic injections of radiotracer and dyes.
Procedure: Endoscopic NIR imaging and gamma probe — Endoscopic near infrared (NIR) imaging of ICG and detection of radiotracer with gamma probe after standard removal of rectal neoplasm.
Procedure: Dissection of sentinel lymph node(s) — Surgical removal of identified lymph nodes in the rectum.

SUMMARY:
The purpose of this study is to develop a technique that allows physicians to identify the first lymph nodes draining from a rectal tumor (the sentinel lymph nodes). Currently, there is no technique used to find these lymph nodes in the rectum during surgery and therefore many patients with rectal cancer need to undergo a total rectal resection. Dyes, tracers, imaging and a gamma probe will be used in this study during a standard minimally invasive transanal endoscopic surgery (TES) to try to locate these lymph nodes. If surgeons are able to locate these lymph nodes they will be removed during surgery. If the technique is successfully developed as a result of this research, it could help patients in the future with early stage rectal cancer by allowing doctors to see if their cancer has spread to the lymph nodes of the rectum without having to undergo a total rectal resection. These patients would then be able to undergo a TES combined with a lymph node dissection to gain more knowledge about the stage of their disease. This knowledge would then be used to determine if and what further treatment is necessary for the patient's rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective transanal endoscopic surgery (TES) at the University of Virginia for rectal neoplasm (polyp with high grade dysplasia, T1N0 tumors < 3cm in the absence of poor pathologic features, patients that refuse radical resection)
* Willing and able to give written informed consent

Exclusion Criteria:

* Patients less than 18 years of age
* Women who are pregnant and/or breastfeeding
* Prisoners
* Unable to give written informed consent
* Patients with any of the following:

  * Allergy to technetium, Spot and/or ICG
  * Allergy to iodides
  * Severe cardiac disease (hospitalization for cardiac disease in the last year, congestive heart failure, abnormal EKG) or renal disease (Creatinine > 2.0 mg/dL)
* Patients with medical contradictions or have potential problems complying with the requirements of the protocol, in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
1st Phase: Detection rate of sentinel lymph node in first 6 patients | Throughout first phase of study, an average of 1 year.
  Data from the first 6 eligible patients will be used to verify feasibility. For this phase, the data need to support a detection rate of at least 50% for the procedure to be considered feasible to move forward with the 2nd phase. The proposed SLNm technique will be declared 'feasible' if at least one SLN is identified per patient. Identification of the SLN in three consecutive patients would provide 80% confidence of successful identification more than 50% of the time. A total sample of size of 6 patients would allow for three refinements in technique if necessary to establish feasibility.
2nd Phase: Detection rate of refined protocol in identifying SLN | Throughout first phase of study, an average of 1.5 years.
  2nd Phase: Sample size is set at 16 eligible patients. For this study, continued investigation of the proposed technique would be of interest if 70-100% of the SLNs are detected. If at least on SLN is detected in 14 of 16 patients, an observed rate of 87.5%, then the lower limit of a one-sided 90% confidence interval is 70%. Thus, detection of at least one SLN in 14 or more patients out of 16 assessed would provide strong preliminary data for the technique (i.e. SLN is detected in at least 70% of patients). If it's assumed, on average, 1.5 SLN could be identified and excised per patient, then with 24 possible SLN, the estimated rate of SLN positive for disease would have an expected half width (or precision of the estimate) of 12-14%.

SECONDARY OUTCOMES:
Size of the SLN according to pathologic analysis | Throughout study, an average of 2.5 years
Location of the SLN according to pathologic analysis | Throughout study, an average of 2.5 years.
Time required for completion of the protocol | Throughout study, an average of 2.5 years.
Number of protocol modifications for procedural and/or technical issues | Throughout study, an average of 2.5 years
Ergonomic optimization of the protocol as measured by operative time | Throughout study, an average of 2.5 years
Ergonomic optimization of the protocol as measured by surgeon satisfaction | Throughout study, an average of 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Traci Hedrick, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States